CLINICAL TRIAL: NCT02428283
Title: The Effect of Scalp Nerve Block on the Emergence Agitation in Children Undergoing Nevus Surgery During Sevoflurane Anesthesia
Brief Title: Scalp Nerve Block on Emergence Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-MED-CT4-14-422
Record Dates: First submitted 2015-04-21; First posted 2015-04-28 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Ropivacaine; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nerve block (Experimental): Scalp nerve block was performed with 0.25% ropivacaine.
  Interventions: Drug: Ropivacaine; Drug: Sevoflurane
- Control (Active Comparator): Remifentanil was administered intravenously.
  Interventions: Drug: Remifentanil; Drug: Sevoflurane

INTERVENTIONS:
Drug: Ropivacaine — 0.25% ropivacaine 2-3 ml was injected around the scalp nerves that are located on the head.
  Arms: Nerve block
Drug: Remifentanil — Remifentanil 1 μg/kg was injected before skin incision.
  Other Names: Ultiva
  Arms: Control
Drug: Sevoflurane — Anesthesia was titrated with sevoflurane, maintaining mean arterial pressure and heart rate within 20% baseline value.

SUMMARY:
Emergence agitation is a common problem in children during recovery from sevoflurane anesthesia. Pain is considered as a cause of postoperative emergence agitation and compounding factor of agitation assessment in children. The purpose of this study was to investigate the effect of scalp nerve block on the emergence agitation in children undergoing nevus surgery during sevoflurane anesthesia.

DETAILED DESCRIPTION:
Forty-four children, 1-7 years old, undergoing nevus surgery on head were enrolled. Anesthesia was induced with thiopental sodium and rocuronium, and maintained with sevoflurane. Patients were randomly assigned two groups: the control group received IV remifentanil 1 μg/kg, and the block group received scalp nerve block with 0.25% ropivacaine 2-3 ml. Time to tracheal extubation, recovery time, hemodynamic change, FLACC score, and Watcha behavior scale for emergence agitation were assessed.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients undergoing general anesthesia for nevus surgery

Exclusion Criteria:

* developmental disorder
* neurologic disorder
* coaguloparthy
* allergy to local anesthetics

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
change of Watcha behavior scale for emergence agitation (4 point) | from immediately after PACU arrival to 10 min, 20 min, and 30 min after arrival

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeongki-do, South Korea